CLINICAL TRIAL: NCT01311011
Title: Phase II Prospective Study of the Clinical Efficacy of Autologous SCT in Patients With Critical Limb Ischemia
Brief Title: Study of the Clinical Efficacy of Autologous SCT in Patients With Critical Limb Ischemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: RAC# 2081-026; RAC# 2081-026
Record Dates: First submitted 2011-03-06; First posted 2011-03-09 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Critical Limb Ischemia
Keywords: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: SCT — SCT

SUMMARY:
Phase II Prospective Study of the Clinical Efficacy of Autologous SCT in patients with Critical Limb Ischemia

DETAILED DESCRIPTION:
Phase II Prospective Study of the Clinical Efficacy of Autologous SCT in patients with Critical Limb Ischemia

ELIGIBILITY:
Inclusion Criteria:

* Patients with Critical Limb Ischemia

Exclusion Criteria:

* Patients with other than Critical Limb Ischemia

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Critical Limb Ischemia
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2008-11

CONTACTS AND LOCATIONS:
Overall Officials: H Al-Zahrani, M.D., Principal Investigator — KFSH & RC
Locations (1):
- Kfsh & Rc, Riyadh, Saudi Arabia